CLINICAL TRIAL: NCT05298345
Title: Descriptive Study of the Family Champions Project
Brief Title: Family Champions Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Anthem Strong Families (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2021/03/36
Record Dates: First submitted 2022-02-28; First posted 2022-03-28 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Fathers; Mothers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Workshop Sessions (Experimental): Participants receive 18 total workshop hours; TYRO Leadership curriculum in 6 2-hour weekly sessions for a subtotal of 12 hours, and Core Communication curriculum in 1-3 sessions for a subtotal of 6 hours.
  Interventions: Other: Family Champions Project Primary Services

INTERVENTIONS:
Other: Family Champions Project Primary Services — Primary Services: participants receive 12 hours of TYRO Leadership curricula, 6 hours of Core Communication curricula.
  Support Services (optional): participants choose from a menu of classes (1-3 hours) at the walk-in mini clinic to meet a variety of self-identified needs.

SUMMARY:
This evaluation uses a formative approach and a descriptive design with repeated measures to assess the efficacy of a Continuous Quality Improvement (CQI) Process to improve services delivered by the Family Champions Project (FCP). The FCP delivers education-based services-TYRO Leadership and Core Communication curricula-with funding from the Office of Family Assistance to low-income fathers and mothers to promote healthy family relationships and economic stability in their households. TYRO Leadership and Core Communication are adapted from the TYRO suite of curricula that were developed by the RIDGE Project, and they are designed to improve the relationships of families affected by the incarceration of a parent and the economic stability of their households. Participants must be at least 18 years of age with a child no older than 24 years and have no open criminal cases (cases can be deferred). Evaluation activities are carried out by Midwest Evaluation and Research (MER) and assess the extent to which our CQI Process is a feasible approach to improve outputs and the outcomes that might be associated with them for an education-based service delivery effort like the FCP.

Specifically, study results from formative evaluation will inform practitioners in the field of HMRE about the viability of using a CQI Process like ours to achieve full implementation and provide some evidence about its capacity to improve outcomes. Formative evaluation not only assesses experiences of the CQI Team and front-line service staff while implementing our CQI Process, but also pays attention to the timing and other specifics of any performance interventions that occur over the 5-year project. As a result, performance interventions present opportunities to conduct a series of mini studies to descriptively evaluate CQI Team efforts to improve implementation of the FCP. Performance trends that improve after an intervention indicate the CQI Team was likely successful to more fully implement outputs which should result in a positive effect on retention rates and, in turn, short term outcomes if we assume a sound theory of change for the FCP is depicted in the logic model.

DETAILED DESCRIPTION:
Efforts to conduct CQI are in the early stages of development in the field of Healthy Marriage and Relationship Education (HMRE). The Office of Family Assistance (OFA) has required HMRE grantees to conduct CQI as part of project activities since funding began for them in 2006. However, HMRE grantees have likely not bought into the CQI Process given the absence of user-friendly conceptual frameworks to guide CQI efforts and empirical evidence to demonstrate they improve implementation of project activities and, in turn, enhance participant outcomes that might be attributed to them.

The CQI Process used in this study was developed by Dr. Theodore C. Jurkiewicz and then enhanced after starting work at MER, and it begins by forming a CQI-Team. The CQI-Team is a collaboration between practitioners with the authority to make implementation decisions about the FCP and evaluators at MER who handle data analyses and reporting.

The CQI Team carries out a multistep plan that is repeated each program year to fully implement FCP educational services over time by using a series of indicators to track performance trends for various outputs from a different perspective in each step. Percentage of target enrollment, percentage of target population that reflect eligibility characteristics, hours of dosage received by participants, response rates to participant surveys that measure outcomes among other indicators and outputs are tracked for monthly and quarterly enrollment cohorts in each program year and presented in CQI Reports that take the perspective associated with each of the steps. The CQI Team discusses findings presented by evaluators for overall performance trends in bi-weekly reports for the 1st step and performance trends by site in quarterly reports presented twice per year for steps 2 and 3. Then, members of the CQI-Team collaborate with front line service staff to develop interventions for any performance trend with an output that seems likely to fall short of standards by the end of the program year. Effects of interventions on outputs are reported by site in step 4.

Ultimately, successful performance interventions designed and implemented by the CQI Team in collaboration with front-line service staff should improve the outputs associated with FCP services over time, and the most immediate impact should be evident in participant retention rates. Interventions that lead to higher enrollment and then improved attendance should lead to a higher incidence of complete program status (active, complete, not in program), which means FCP services are being delivered to more participants in larger doses. Larger doses of services delivered to participants after performance interventions which means the CQI Team is facilitating progress to meet performance standards because participants receive the amounts of FCP services intended for them.

What is more, higher retention rates over time should lead to improved short-term outcomes for participants. Participants who receive larger doses of FCP services after performance interventions should acquire more knowledge in educational sessions than those who receive smaller doses. However, rigorous measures of participant knowledge are not available because it was not possible to get full access to proprietary curricula to develop them. Consequently, participant attitudinal changes will be the only focus for measuring short-term outcomes in this study. Attitudes change more quickly in healthy and productive ways after merely exposing participants to new ways of thinking about parenting, handling finances, or accessing employment with curriculum content in the FCP.

Finally, FCP services cannot determine participant outcomes but only contribute to them amongst a host of other factors, which makes it difficult for a descriptive study to link behavioral change to CQI efforts. Healthier and more productive behaviors take time to emerge, develop, and hopefully replace old behaviors because they are subject to a host of other influences on FCP participants. What is more, low-income individuals in the FCP target population, especially those who are parents, experience changing life circumstances more often than those from wealthier households that make them more vulnerable to a host of risk-related factors, such as unstable employment, tenuous housing situations, or limited sources of support that are available from family and friends. Changing life circumstances for low-income individuals make it more difficult for FCP services to have a positive, lasting impact on their behavior.

In sum, immediate effects of successful performance interventions that result from the CQI Process should be evident in retention rates for FCP services over time because they are being delivered to more participants in larger doses, as indicated by more hours of attendance in TYRO Leadership and Core Communication workshops and higher workshop completion rates. Higher retention rates mean more participants acquire more knowledge from curriculum content to influence their attitudes about partner relationships.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and older)
* Parent
* No open criminal cases (or deferred)

Exclusion Criteria:

* Minor (under the age of 18)
* Not a parent
* Has an open criminal case (or not deferred)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1111 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation & Research
Locations (1):
- Anthem Strong Families, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Workshop Sessions: Participants receive 18 total workshop hours; TYRO Leadership curriculum in 6 2-hour weekly sessions for a subtotal of 12 hours, and Core Communication curriculum in 1-3 sessions for a subtotal of 6 hours.
  Family Champions Project Primary Services: Primary Services: participants receive 12 hours of TYRO Leadership curricula, 6 hours of Core Communication curricula.
  Support Services (optional): participants choose from a menu of classes (1-3 hours) at the walk-in mini clinic to meet a variety of self-identified needs.
Period: Overall Study
Arm/Group | Primary Workshop Sessions
Started | 1111
Completed | 1111
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary Workshop Sessions
Number analyzed (Participants) | 1111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1088
  >=65 years | 23
Age, Continuous [Mean (Full Range); unit: years] | 39.93 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 944
  Male | 167
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 44
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 11
  Black or African American | 211
  White | 667
  More than one race | 167
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure 1: Retention Rates Among Participants
Description: Do FCP participants exhibit higher retention rates (i.e., completion %) after cycles of CQI?
  • Measured by program status (% active, complete, or not in program) as recorded on the nFORM online data collection system whose use is required by the funder to track programmatic data, such as enrollment and participation levels.
  Count of participants who dropped out before CQI efforts began was obtained Count of participants who dropped out after CQI efforts began was obtained Count of participant completions before CQI efforts began was obtained Count of participant completions after CQI efforts began was obtained
Time Frame: through study completion, an average of six weeks
Population: These numbers are inconsistent with numbers provided in the rows in the Participant Flow module due to the number of participants who were included in the sample of the study (which is much smaller than the overall number enrolled). This is due to the study only looking at a portion of the study where this process was implemented.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Workshop Sessions
Number analyzed (Participants) | 187
Participants
  # of dropouts pre intervention | 20
  # of dropouts post-intervention | 13
  # of completions pre intervention | 76
  # of completions post-intervention | 78

2. Secondary Outcome: Secondary Outcome Measure 1: Partner Relationship Attitudes
Description: Do FCP participants exhibit healthier partner relationship attitudes after enrolling in the program?
  * 5 survey items measure the reported frequency of agreement with healthy partner relationship attitudes on a 4-point scale (1 'Strongly Agree', 2 'Agree', 3 'Disagree', 4, 'Strongly Disagree', NA 'Not Applicable').
  * Lower scores on all items are positive (ex. - I want to grow old with my partner.)
  The 5 items are measured as a construct. All items are added together and divided by 5 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: pre to post completion which is 6 weeks longs
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Workshop Sessions
Number analyzed (Participants) | 485
score on a scale
  mean at baseline | 3.22 (.707)
  mean at follow-up | 3.50 (.611)

ADVERSE EVENTS:
Time Frame: up to 10 weeks
Description: The definitions of adverse events do not differ from the clinicaltrials.gov definitions.
Arm/Group | Primary Workshop Sessions
All-Cause Mortality (participants affected / at risk) | 0/1111
Serious Adverse Events (participants affected / at risk) | 0/1111
Other Adverse Events (participants affected / at risk) | 0/1111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT05298345/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT05298345/SAP_001.pdf